CLINICAL TRIAL: NCT02685137
Title: A Multicenter Study to Evaluate the Efficacy and Safety of Tin Mesoporphyrin (Stannsoporfin) to Reduce the Need for Phototherapy in Term and Near Term Infants.
Brief Title: Efficacy and Safety of Stannsoporfin in Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 64,185-01-3W
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2018-06

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: Kernicterus; Neonatal Jaundice; Newborn Jaundice; Hyperbilirubinemia; Stannsoporfin
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Kernicterus; Jaundice, Neonatal; Hyperbilirubinemia | interventions — tin mesoporphyrin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active drug-Stannsoporfin (Experimental): Stannsoporfin, single dose 4.5mg/kg administered Intramuscular (parental injection in the thigh) for treatment of jaundice
  20 mg/mL 1.5 mL/vial
  Interventions: Drug: stannsoporfin
- Reference Therapy-Sham (Sham Comparator): Sham Injection, no injection followed by a Band-Aid to thigh
  Interventions: Other: Sham Injection

INTERVENTIONS:
Drug: stannsoporfin — Intramuscular injection of stannsoporfin to treat jaundice.
  Arms: Active drug-Stannsoporfin
Other: Sham Injection — nothing
  Arms: Reference Therapy-Sham

SUMMARY:
This is a multi-center, randomized, sham injection-controlled (placebo) masked trial of a single intramuscular injection of Stannsoporfin compared to "sham" (placebo) in healthy term and near-term newborns admitted to the well-baby nursery and enrolled with "intention to treat".

DETAILED DESCRIPTION:
For purposes of analysis, 2 patient populations are defined. One population consists of those babies who did not develop severe hyperbilirubinemia (TSB <9 mg/dL) during the first 36 hours of age. This population is referred to as the untreated population of screened but not randomized patients. The second population of babies was defined as those infants who develop severe hyperbilirubinemia. These infants were randomized to treatment with either stannsoporfin or the sham injection and will be the focus of the efficacy and safety analysis. This population was referred to as the treated population.

The treated population was used for the efficacy and safety analysis. These infants were randomized to either stannsoporfin or the sham injection treatment group.

ELIGIBILITY:
Patients were enrolled who meet the following criteria:

1. The infant's family may be approached at anytime from 6 hours after birth onward to discuss the possibility of enrollment. However, Informed Consent may not be signed until the baby is between 12 and 36 hours of age.
2. Consent may be obtained as soon as possible after 12 hours of age, when the baby enters the well-baby nursery.
3. An infant may be included if the mother has received, or the baby is receiving, antibiotics and the infant is asymptomatic. For example, the baby has no signs of cardiorespiratory distress and is feeding well. Symptomatic infants are excluded (see Exclusions, below).
4. Born at the study hospital site and admitted to the well-baby nursery or admitted to the intensive-care nursery for <12 hours for post delivery observation (delayed transition, temperature or dextrose instability, meconium staining and/or parental concern).
5. All babies on oral feeding with stable cardiorespiratory status and deemed "healthy" upon clinical examination, with normal perfusion as defined by capillary filling of the fingernail.
6. Term neonate (≥38 weeks of completed gestation), OR
7. Near-term neonate (>36<38 weeks of completed gestation; >2,000g birth weight), OR
8. Near-term neonate (>35<38 weeks of completed gestation; >2,500g birth weight)
9. Care provided (primarily) in the well-baby nursery population;
10. Absence of concurrent cardiorespiratory distress, sepsis, major congenital anomalies or need for care in an intensive care nursery;
11. Not participating in another concurrent unrelated study.

Exclusion Criteria

The study enrolled patients who did not have any of the following exclusion criteria:

1. Any condition that in the opinion of the investigator would make the subject unsuitable for the study.
2. Infants receiving antibiotics who are also symptomatic are excluded. For example, a baby who is feeding poorly or is in cardiorespiratory distress is excluded.
3. Mother has received phenobarbital in past 30 days.

Ages: 12 Hours to 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2002-05-01 (Actual); Primary Completion 2003-03-16 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Need for Phototherapy | 30 days
  proportion of cases which need phototherapy in the treated population

SECONDARY OUTCOMES:
hyperbilirubinemia | 12 hrs
  Change in serum bilirubin values

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States